CLINICAL TRIAL: NCT03036007
Title: Physiotherapy After Anterior Cervical Spine Surgery for Cervical Disc Disease. A Prospective Randomised Study to Compare Internet-based Neck-specific Exercise With Prescribed Physical Activity
Brief Title: Physiotherapy After Anterior Cervical Spine Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, PT, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016 / 283-31
Record Dates: First submitted 2017-01-18; First posted 2017-01-30 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cervical Disc Disease; Radiculopathy, Cervical
Keywords: Spine, Disc, Neck pain, Rehabilitation, Exercise Therapy, Internet
MeSH Terms: conditions — Radiculopathy; Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescribed Physical Activity (Active Comparator): General physical exercises combined with 3 visits at a physiotherapy clinic (plus an additional first visit), exercises mainly performed outside the health care system during 12 weeks.
  Interventions: Other: Prescribed Physical Activity
- Exercises with Internet support (Experimental): Neck-specific exercises with Internet support combined with 3 visits at a physiotherapy clinic (plus an additional first visit), exercises mainly performed outside the health care system during 12 weeks.
  Interventions: Other: Exercises with Internet support

INTERVENTIONS:
Other: Prescribed Physical Activity — General physical activity prescribed by a physiotherapist
  Arms: Prescribed Physical Activity
Other: Exercises with Internet support — Neck-specific exercise with Internet support
  Arms: Exercises with Internet support

SUMMARY:
Background: Patients suffering residual disability after anterior decompression and fusion (ACDF) surgery for cervical disc disease may be prescribed physical activity (PPA) or neck-specific exercises (NSE). Currently, we lack data for the success of either approach. There is also a knowledge-gap concerning the use of internet-based care for chronic neck pain, inclusive of cervical disc disease. The scarcity of these data, and the high proportion of patients with various degrees of incapacity following ACDF, warrants increased efforts to investigate and improve cost-effective rehabilitation.

Objective: To investigate the effectiveness of a structured, internet-based NSE program, versus PPA following ACDF surgery.

Methods: This is a prospective, randomised, experimental, longitudinal multicentre study, that includes 140 patients with residual disability (≥30% on the Neck Disability Index; NDI) following ACDF for radiculopathy due to cervical disc disease. Patient recruitment occurs following attendance at routine clinical appointments, scheduled for 3-months post-surgery. Patients are then randomised to one of two groups (70 patients/group), scheduled for a 3-month treatment of either internet-based NSE or PPA. Questionnaires on background data, pain and discomfort, physical and mental capacity, satisfaction with care, and health and workplace factors are completed, with physical measurements of neck-related function performed by independent test leaders blinded to randomisation. Measurements are performed at inclusion, after the 3-month treatments (end of treatment), and at a 2-year follow-up. Radiography will be completed at the 2-year follow-up. Preoperative data will be collected from the Swedish Spine Registry (Swespine). Data on healthcare consumption, drug use, and sick leave will be requested from the relevant national registers.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether internet-based, structured NSE, differs from PPA after surgery for cervical disc disease, in relation to function, pain, work capacity, health-related quality of life, satisfaction with care, and cost effectiveness.

The hypothesis is that internet-based NSE will be superior in terms of outcome measures to PPA. This assumption, based on an earlier study of patients with chronic WAD, remains untested for individuals with residual disability following ACDF. The project is expected to lead to improved care, well-being, and patient satisfaction, and, as a result, a reduced societal burden.

Design This is a prospective, randomised, experimental longitudinal multicentre study, with a two-year follow-up. Questionnaires are distributed and physical measurements taken at baseline, at the end of treatment (3 months after enrolment), and after 2 years. Preoperative data is collected from Swespine. Patients are recruited from the surgical unit following regular follow-up visits to the physiotherapist/surgeon at approximately 3 months postoperatively.

Should the study criteria be met, and after the receipt of written and oral informed consent, the patient completes a questionnaire and undergoes physical measurements of neck-related function. The patient is then randomised (computerised block randomisation list compiled by statisticians) to one of two groups for 3 months of treatment with a) internet-based NSE with 3 visits to the physiotherapist or b) PPA with 3 visits to the physiotherapist. In addition, and prior to treatment, patients in both groups are examined by a physiotherapist, in accordance with Swedish law.

The test leader is a physiotherapist at the surgical unit who is not involved in study treatment and is blinded to the randomisation groups. Qualified clinicians will perform X-rays and (potentially) ultrasound registration. Following randomization the results will be put into an opaque envelope that contains the name of the patient and their randomisation group, which is sent to the physiotherapy outpatient care clinic. Questionnaires and tests of physical neck-related function are conducted at baseline (before randomisation), after 3 months (when the treatment ends), and after 2 years. Participant physiotherapists will be provided oral, written, and practical training, and are able to consult project managers at any time. Exercise diaries and the number of care contacts will be recorded for both groups.

Study criteria

Inclusion criteria for each surgical department:

• Record data in Swespine

Inclusion criteria for surgery:

* Cervical disc disease, confirmed by MRI data compatible with clinical findings (neurological examination performed by neck surgeon i.e. neurosurgeon/orthopaedic surgeon) that show nerve root compression in the cervical spine.
* Radiculopathy with pain in one or both arms, with or without sensory and/or motor deficit
* At least 3 months of persistent arm pain

Inclusion criteria for the study:

* ACDF due to cervical disc disease (disc herniation with or without osteophytes, or stenosis caused by osteophytes) in one or two segmental levels
* Age 18-75 years
* Residual disability (approximately) 3 months after surgery (at the re-visit to the surgeon/ physiotherapist at the neurosurgery/ neuroorthopedic clinic) in terms of the Neck Disability Index (NDI ≥30%).
* Access to a computer/tablet/smartphone and the Internet
* Motivated to exercise

Exclusion criteria:

* Myelopathy
* Previous fracture or dislocation of the cervical spine
* Malignancy or benign spinal tumour (e.g. neuromas)
* Spinal infection, ongoing post-operative infection, or previous spondylodiscitis
* Previous cervical spine surgery
* Factors that are contraindicated for study participation or which hinder treatment or follow-up because of systemic disease, physical or mental illness, injury, inconvenience, or postoperative complications.
* Known alcohol/drug abuse
* Lack of ability to write/comprehend/or express oneself in the Swedish language

Intervention Internet-based neck-specific exercise (NSE) Participants will be provided with an explanation and justification for their exercise. Training includes exercises to activate the deep neck muscles (initially daily), continuing with endurance training of the neck and shoulder muscles (3 times/week). Exercise will be tailored to the individual's physical condition, and then scaled up progressively in terms of severity and dose. Participants will undertake three visits to the physiotherapist, where the exercises will be introduced and repeated, in order to establish and control patient comprehension. The exercise is completed with the help of internet support outside of the healthcare system, which can be accessed anywhere, but most probably at home. Photos and videos of the exercises, information, and answers to frequently asked questions are available on the internet-support platform. Patients can contact a physiotherapist by e-mail if necessary. Three visits to the physiotherapist are provided in addition to a mandatory first visit (for new clinical investigations as required by Swedish law). At the end of the treatment period, the patients are encouraged to continue practicing the exercises on their own.

Prescribed physical activity (PPA) The training consists of general, physical, land-based activity (3 times/week). The aim is to find a physical activity outside of the care unit that suits the individual, based on their specific needs and problems. The goal is that the individual should increase their overall level of physical activity, and that that activity is performed as part of a self-care/wellness routine. This may involve activities that can be performed at home, such as walking according to a set schedule, home exercises given by a physiotherapist (not neck-specific training), and aerobic classes etc. To increase compliance, a simple motivational interview is performed before the PPA schedule is provided, which can occur during the same session or at a separate visit, should the physiotherapist and patient prefer. Patients are advised to contact the physiotherapist should their prescribed activity fail to work so that another activity can be identified. Three visits to the physiotherapist are provided in addition to a mandatory first visit (for new clinical investigations as required by Swedish law), with the patient encouraged to continue practicing on their own at the end of the treatment period.

Sample size calculation and statistics Seventy participants per group (i.e. a total of 140 patients) are required. Sample size calculations (conducted by statisticians) are based on the primary outcome measure of Neck Disability Index (NDI). In order to detect a clinically relevant improvement of 10 NDI points, 70 participants per group are needed (assuming 80% power, and a level of significance of 5%). This calculation is based on group differences recorded in previous studies. These include a study in which individuals with chronic whiplash-associated injuries were offered training, as well as a study investigating the benefits of surgery over and above physical therapy for cervical disc disease.

As we lack any studies on rehabilitation for patients with disability after ACDF, this calculation remains hypothetical and our sample size may need to be adjusted after the first 30 people (15/group) have completed the 3-month follow-up. This number can also be adjusted in the event of participants dropping-out, such that at least 70 individuals per group complete the intervention. Data will be analysed using an intention-to-treat approach. Alternative analyses (sub-group analyses) will be carried out where the degree of implementation of treatment (compliance) is taken into account, as well as sex, dizziness, headaches, neurological findings, and the number of segmental levels operated on. Analyses will be performed using parametric or non-parametric statistics, depending on the type of data, in consultation with statisticians as appropriate.

Ultrasound registrations, electromyography, Magnetic Resonance Imaging and kinesthesia may be done on a sub-group of participants to investigate neck muscle structure and function. Interviews may be done on a sub-group of individuals regarding their function, experiences and opinions.

Ethical considerations This study was approved by the Regional Ethical Review Board in Linköping Ref: 2016 / 283-31. The scientists are independent with no commercial ties. Patients are recruited after providing informed consent. Patient data are presented at the group level such that no connection to any individual can be made. All data are anonymised when reported, and subject to the Official Secrets Health Acts. The test leaders are independent and blinded for randomisation. Exercises, both general and neck-specific, have been used extensively in clinical practice and we anticipate no harm from their implementation other than a risk of muscle soreness. Any important harms or unintended effects in each group will be collected by the test leaders. All questionnaires and test materials are encoded by the research group, with code lists stored in locked, fireproof file cabinets, housed at the university in a room with controlled (card-based) access. Only individuals in receipt of a unique website address posted by the researchers can access the program; patients can neither communicate with each other nor with caregivers via the program.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for each surgical department:

• Record data in Swespine

Inclusion criteria for surgery:

* Cervical disc disease, confirmed by MRI data compatible with clinical findings (neurological examination performed by neck surgeon i.e. neurosurgeon/orthopaedic surgeon) that show nerve root compression in the cervical spine.
* Radiculopathy with pain in one or both arms, with or without sensory and/or motor deficit
* At least 3 months of persistent arm pain

Inclusion criteria for the study:

* ACDF due to cervical disc disease (disc herniation with or without osteophytes, or stenosis caused by osteophytes) in one or two segmental levels
* Aged 18-75 years
* Residual disability (approximately) 3 months after surgery (at the re-visit to the surgeon/ physiotherapist at the neurosurgery/ neuroorthopedic clinic) in terms of the Neck Disability Index (NDI ≥30%).
* Access to a computer/tablet/smartphone and the Internet
* Motivated to exercise

Exclusion Criteria:

Exclusion criteria:

* Myelopathy
* Previous fracture or dislocation of the cervical spine
* Malignancy or benign spinal tumour (e.g. neuromas)
* Spinal infection, ongoing post-operative infection, or previous spondylodiscitis
* Previous cervical spine surgery
* Factors that are contraindicated for study participation or which hinder treatment or follow-up because of systemic disease, physical or mental illness, injury, inconvenience, or postoperative complications.
* Known alcohol/drug abuse
* Lack of ability to write/comprehend/or express oneself in the Swedish language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up. Preoperative data from the Swespine register
  Self-reported neck-specific function

SECONDARY OUTCOMES:
Pain intensities of the neck, arm, and head, measured using the Visual Analogue Scale (VAS 0-100 mm). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up. Pre-operative data from the Swespine register
  Pain intensity VAS
Pain intensities for the neck and arm will be assessed and registered using the Numeric Rating Scale (NRS) 0-10 scale in accordance with the Swespine registry | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Pain intensity NRS
Distribution of pain by a Pain Drawing assessed with images | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  painful areas are shaded on a human body image
Use of pain medications | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Use of pain medications
Modified Odom | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  global outcomes of the intervention
Dizziness/balance by the Dizziness Handicap Inventory (DHI) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Self-reported dizziness
Headache questions by VAS and the Headache Handicap Inventory (HIT-6) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Impact of headache
Disaster thoughts measured by the Pain Catastrophising Scale (PCS). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Disaster thoughts
Confidence in ability measured by the Self-Efficacy Scale (SES). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Confidence in ability
Patient Specific Functional Scale (PSFS). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Estimation of neck-specific function related to participants' chosen activities (daily function, work, spare time
Fear Avoidance Beliefs Questionnaire (FABQ). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Operating fear
Hospital Anxiety and Depression Scale (HAD). | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Self-reported anxiety and depression
Health related quality of life measured by the EuroQuol five dimensions (EQ-5D) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Health related quality of life
Work Ability Index (WAI), short form | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Self-rated work ability
Requirements - effort support in the workplace: Effort Reward Imbalance (ERI) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  effort and support in the workplace
Ergonomics questions and how work is perceived | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Work ergonomics
Sickness presence measured by the Stanford preseenteism scale | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Sickness presence at work
Swedish Standard Classification of Occupations (SSY) code | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Classification of Occupations
Patient Enablement Instrument (PEI) questionnaire | Follow-up at 3 months (the end of treatment) and 24 months follow-up
  Patient Enablement
Satisfaction with symptoms measured by the Cherkin symptom satisfaction scale | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Satisfaction with symptoms
Level of physical activity score, a combination of 2 questions (everyday physical activity and exercise/sport/open-air activity) to a combined 4-point score | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Physical activity
Health-care consumption, number of visits | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Health-care consumption
Consumption of analgesic drugs prescribed through the drug registry | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Consumption of analgesic drugs
Frequency of pain | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Frequency of pain
Sick-leave registration, number of days and episodes | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Sick-leave registration
Neck movement measured using the cervical range of motion device (CROM) in degrees | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Active range of motion
Endurance in the dorsal and ventral neck muscles, measured in seconds | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Neck muscle endurance
Sensorimotor control of ventral neck muscles, in the supine position, with stabilizer (mm HG) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Sensorimotor control
Neurology, clinical judgement yes/no | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Neurology, such as reflexes, sensibility, muscle weakness and neural tension test. The results of the neurological examination gives an overall clinical judgement if segmental neurological findings is present and which cervical segmental level/ - is involved,
Hand strength measured with a hand dynamometer (Jamar) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Hand strength
Standing on one leg with eyes closed (Solec test) | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Static balance
Conventional radiography, with side views taken during neutral positioning and dynamic flexion/extension | Occurs routinely in the clinic for visits 3 months after surgery. Additional X-rays will be taken at the 2-year follow up to
  Examination of implants, the degree of mobility of operated segments, subsidence and fusion
Register data for care use. To measure/monitor care use | Change from baseline to 3 months (the end of treatment) and 24 months follow-up
  Care use
MRI may be measured in a sub-group | Change from baseline to 3 months follow-up
  Neck muscle structure and maybe function
Ultrasound registrations may be measured in a sub-group, deformation and deformation rate | Change from baseline to 3 months follow-up
  Neck muscle function
Global rating of change scale | Change from baseline to 3 and 24 months follow-ups, measured at follow-ups
  Overall change because of the treatment

OTHER OUTCOMES:
Background data such as age and gender | Baseline
  Background data such as age, gender, living circumstances and earlier care

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Professor, Principal Investigator — Dep. Medical and Health Sciences, Physiotherapy, Linköping University, Linköping, Sweden
Locations (1):
- Anneli Peolsson, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peolsson A, Peterson G, Hermansen A, Ludvigsson ML, Dedering A, Lofgren H. Physiotherapy after anterior cervical spine surgery for cervical disc disease: study protocol of a prospective randomised study to compare internet-based neck-specific exercise with prescribed physical activity. BMJ Open. 2019 Feb 19;9(2):e027387. doi: 10.1136/bmjopen-2018-027387. PMID 30782952